CLINICAL TRIAL: NCT00902512
Title: Relative Bioavailability Of Two Sildenafil 100mg Oral Tablet Formulations In Healthy Volunteers Under Fasting Conditions.
Brief Title: Study Of Bioavailability Of Two Sildenafil 100mg Oral Tablet Formulations
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Collaborators: Investigacion Farmacologica y Biofarmaceutica, S.A. de C.V. (Other)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: A1481267
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Healthy Males
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Treatment A (Active Comparator): Viagra® 100 mg tablet, administered with water
  Interventions: Drug: Treatment A; Drug: Blood samples for the analysis of sildenafil in plasma
- Treatment B (Active Comparator): Sildenafil 100 mg CT administered with water
  Interventions: Drug: Treatment B; Other: Blood samples for the analysis of sildenafil in plasma
- Treatment C (Active Comparator): Sildenafil 100 mg CT administered without water
  Interventions: Drug: Treatment C; Other: Blood samples for the analysis of sildenafil in plasma

INTERVENTIONS:
Drug: Treatment A — Viagra® 100 mg tablet, administered with water single dose
  Arms: Treatment A
Drug: Blood samples for the analysis of sildenafil in plasma — Blood samples for the analysis of sildenafil in plasma
  Arms: Treatment A
Drug: Treatment B — Sildenafil 100 mg CT administered with water single dose
  Arms: Treatment B
Other: Blood samples for the analysis of sildenafil in plasma — Blood samples for the analysis of sildenafil in plasma
  Arms: Treatment B
Drug: Treatment C — Sildenafil 100 mg CT administered without water single dose
  Arms: Treatment C
Other: Blood samples for the analysis of sildenafil in plasma — Blood samples for the analysis of sildenafil in plasma
  Arms: Treatment C

SUMMARY:
the pharmacokinetics of sildenafil following single doses of sildenafil CT administered with and without water is similar relative to the conventional oral tablet of sildenafil administered with water.

ELIGIBILITY:
Inclusion Criteria:

* Only healthy male volunteers in the 18-40 age range will be included.
* At the selection visit allowed normal range for vital signs will be: Blood pressure (with the subject sitting down) 90-130mm Hg systolic and 60-90
* The volunteers' health condition will be determined from their complete clinical history by doctors at the clinical research site and lab test results by certified clinical laboratories mm Hg diastolic, heart rate 55-100 bpm , respiratory rate 14-20 respirations per minute.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at time of dosing) disease or clinical findings at Screening.
* Treatment with a PDE-5 inhibitor within the 4 days preceding the first dose of study medication
* History of hypersensitivity to sildenafil citrate or any components of its formulations

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2009-04; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
AUC0-T and Cmax of sildenafil | 28 days

SECONDARY OUTCOMES:
AUC0-inf of sildenafil | 28 days
Tmax and half-life of sildenafil | 28 days
Adverse events and vital signs | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Col. Arenal Tepepan, Mexico City, Mexico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481267&StudyName=Study%20Of%20Bioavailability%20Of%20Two%20Sildenafil%20100mg%20Oral%20Tablet%20Formulations%0A